CLINICAL TRIAL: NCT03176511
Title: Novel Dual-Task Balance Challenge to Prevent Falls in Older Adults
Brief Title: Fall Prevention in Older Adults Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG2017-13
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2017-05

CONDITIONS: Accidental Fall; Postural Balance
Keywords: older adults; dual task; A Matter of Balance

STUDY DESIGN:
Intervention Model Description: The proposed pilot study will employ a single-blind, two-group randomized clinical trial. We will randomly assign 24 community-dwelling older adults (≥ 60 years) from an underserved population who are at high fall risk to either: A.) 4-week MOB+DTBC intervention, or B.) 4-week MOB only intervention (n=12/group).
Who Masked: Outcomes Assessor
Masking Description: As with any active intervention, participants will know their group assignment and double-blinding is not possible. Of note, our primary outcome measures are objective and require post-processing, thus study staff collecting the data will be "blinded" to participant results. Further, our bio-engineer post-processor will be blinded to study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOB+DTBC Group (Experimental): A Matter of Balance plus Dual-Task Balance Challenge Group. Standardized MOB classes twice/week for 4 weeks, plus 15 minutes of DTBC each class. Each class is 2 hours 15 minutes.
  Interventions: Behavioral: A Matter of Balance plus Dual-Task Balance Challenge Group
- MOB Group (Active Comparator): A Matter of Balance Group. Standardized MOB classes twice/week for 4 weeks, plus 15 minutes of social time each class. Each class is 2 hours 15 minutes.
  Interventions: Behavioral: A Matter of Balance Group

INTERVENTIONS:
Behavioral: A Matter of Balance plus Dual-Task Balance Challenge Group — Participants will receive the standard MOB classes, along with a 15-min DTBC each class, i.e., right and left foot ankle-reaching to three differently colored markers. Three colored dots are placed on the ground in an arc, using different colored stick-on dots. A chair can be placed in front of the color pattern, as needed for safety.
  Other Names: MOB+DTBC Group
  Arms: MOB+DTBC Group
Behavioral: A Matter of Balance Group — Participants will receive the standard MOB class, taught by a certified MOB, using course materials developed by MaineHealth's Partnering for Healthy Aging (http://www.mainehealth.org/pfha).
  Other Names: MOB Group
  Arms: MOB Group

SUMMARY:
Poor balance is one of the major risk factors for falling in older adults. A Matter of Balance (MOB) is one of the most commonly used fall prevention programs nationally. Despite its name, MOB focuses on managing concerns about falling, and does not include a balance component. We are testing to see if adding a dual-task balance component (balance and mental thinking) to MOB can improve balance and walking better, than MOB only.

DETAILED DESCRIPTION:
Fall prevention interventions among community-dwelling older adults are essential. A Matter of Balance (MOB) is one of the most commonly used community-based fall prevention interventions nationally, and is considered the 'fall prevention standard of care'. MOB programs are targeted to reduce the fear of falling and promote physical activity among all older community-dwelling adults. While evidence indicates that the MOB program leads to small, sustained decreases in older adults' perceived fear of falling, there is no evidence of objectively measured balance and gait. Despite its name, MOB focuses on cognitive restructuring to manage concerns about falling, and does not include a balance component. Among community-dwelling older adults, both intact balance and concomitant attention ("dual-tasking") are essential to prevent falls, and dual-task balance components are now requisite per evidence-based fall prevention intervention guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults from all sex/gender and racial/ethnic groups, aged ≥ 60 years, at high fall risk (FRQ=Fall Risk Questionnaire score > 4), who live in the greater Tucson, AZ area.

Exclusion Criteria:

* Older adults currently attending MOB or other fall prevention classes (e.g. Fall Proof), having a severe mobility disorder (e.g., unable to walk 15 feet with an assistive device), severe visual or hearing impairment, non-English speaking, lack of decision-making capacity, unable to provide informed consent, serious psychiatric disorder (e.g., schizophrenia), moderately-severe depression (PHQ-9=Patient Health Questionnaire ≥ 15), cognitive impairment (MMSE=Mini-Mental Status Exam ≤ 23), or serious medical condition (e.g., cancer treatments).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Balance | Data will be collected at baseline and post-intervention at 4 weeks.
  Balance will be assessed using LEGSys™ (Locomotion Evaluation and Gait System, BioSensics LLC) wearable technology. This system uses five sensors attached to right and left anterior shins, right and left anterior thighs, and to the posterior lower back. Balance measures will include changes in sway of ankle, hip, and center of mass (COM) in both mediolateral (ML) and anterior/posterior (AP) directions while standing, with feet parallel and in semi-tandem positions, during eyes-open (EO) and eyes-closed (EC) conditions (30 seconds/test).

SECONDARY OUTCOMES:
Gait | Data will be collected at baseline and post-intervention at 4 weeks.
  Gait will be assessed over a distance of 20 meters using the LEGSys™ wearable technology. The system estimates spatiotemporal gait parameters including velocity, stride length, stride time, double support, single support, and stride-to-stride variability, and gait initiation. COM range of motion during walking will be calculated based on the data from the sensor attached to the lower back. Gait will be assessed under usual and maximal walking speeds.
Fear of Falling | Data will be collected at baseline and post-intervention at 4 weeks.
  Fear of Falling is defined as concerns about falling. The Falls Efficacy Scale International (FES-I) is a self-report measure that assesses concerns about falling for 16 commonly performed activities at home and in community settings (e.g. get in/out of chair, walk in crowded places).
3-month incident Fall Rates | Data will be collected post-intervention at months 1, 2 and 3.
  Participants will be provided with 3 monthly fall calendars and asked to mark it daily (X=no fall, F=Fall) and record details of any fall injury/hospitalization on the back of the monthly sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E Taylor-Piliae, PhD, Principal Investigator — University of Arizona
Locations (1):
- El Rio Community Health Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.